CLINICAL TRIAL: NCT01733979
Title: Efficacy and Safety of Heme-Iron Polypeptide on Improvement of Anemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Wan Chae, Principal Investigator, Clinical Trial Center for Functional Foods, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ABI- IDA-HIPk
Record Dates: First submitted 2012-11-20; First posted 2012-11-27 (Estimated); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — Nonheme Iron Proteins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Heme-Iron Polypeptide (Experimental)
  Interventions: Dietary Supplement: Heme-Iron Polypeptide
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Heme-Iron (Active Comparator)
  Interventions: Dietary Supplement: Heme-Iron
- Organic Iron (Active Comparator)
  Interventions: Dietary Supplement: Organic Iron

INTERVENTIONS:
Dietary Supplement: Heme-Iron Polypeptide — Heme-Iron Polypeptide (1g/day)
  Arms: Heme-Iron Polypeptide
Dietary Supplement: Placebo — Placebo (1g/day)
  Arms: Placebo
Dietary Supplement: Heme-Iron — Heme-Iron (1g/day)
  Arms: Heme-Iron
Dietary Supplement: Organic Iron — Organic Iron (1g/day)
  Arms: Organic Iron

SUMMARY:
The investigators performed a 4-week, randomized, double-blind, placebo-controlled human trial to evaluate the efficacy and safety of Heme-Iron Polypeptide on Improvement of Anemia. The investigators measured Improvement of Anemia parameters , including hemoglobin, transferrin saturation, serum iron, and ferritin, and monitored their blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 19-60 years old
* Hemoglobin concentration less than 13g/dL(men), 12g/dL(women)
* Able to give informed consent

Exclusion Criteria:

* Allergic or hypersensitive to any of the ingredients in the test products
* History of reaction to any of the test products or of gastrointestinal diseases such as Crohn's disease or gastrointestinal surgery
* Participation in any other clinical trials within past 2 months
* History of alcohol or substance abuse
* Laboratory test, medical or psychological conditions deemed by the investigators to interfere with successful participation in the study
* Pregnant or lactating women etc.

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2012-02-07 (Actual); Primary Completion 2012-11-14 (Actual); Study Completion 2012-11-14 (Actual)

PRIMARY OUTCOMES:
Changes in hemoglobin | 4 weeks
  Hemoglobin was measured in study visit 1(0 week) and visit 5(4 week).
Changes in transferrin saturation | 4 weeks
  Transferrin saturation was measured in study visit 1(0 week) and visit 5(4 week).

SECONDARY OUTCOMES:
Changes in serum iron | 4 weeks
  Serum iron was measured in study visit 1(0 week) and visit 5(4 week).
Changes in ferritin | 4 weeks
  Ferritin was measured in study visit 1(0 week) and visit 5(4 week).

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Center for Functional Foods; Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea